CLINICAL TRIAL: NCT04449276
Title: COVID-19: A Phase 1, Partially Blind, Placebo-controlled, Dose Escalation, First-in-human, Clinical Trial to Evaluate the Safety, Reactogenicity and Immunogenicity After 1 and 2 Doses of the Investigational SARS-CoV-2 mRNA Vaccine CVnCoV Administered Intramuscularly in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Vaccine CVnCoV in Healthy Adults for COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CureVac (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: CV-NCOV-001; 2020-001286-36 (EudraCT Number)
Record Dates: First submitted 2020-06-18; First posted 2020-06-26 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2022-04

CONDITIONS: Severe Acute Respiratory Syndrome; Coronavirus; SARS-CoV-2; COVID-19
Keywords: Safety; Reactogenicity; Immunogenicity; Vaccine; CEPI
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections; COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the initial part of the dose escalation, participants will be enrolled in sentinel groups in an open manner. In the second part, participants will be enrolled in placebo-controlled groups in an observer-blind manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation CVnCoV (Experimental): Participants will be vaccinated with CVnCoV at escalating dose levels on Day 1 and Day 29. Safety data will inform the decision to continue enrolling at the current dose level, or to proceed to dose escalation. Initially, dose levels of 2, 4 and 8 μg will be evaluated.
  Dose levels of 2, 4, 6, 8 and 12µg will be evaluated with potential increase to dose levels up to 20 μg.
  Interventions: Biological: CVnCoV Vaccine
- Dose Escalation Placebo (Placebo Comparator): Participants will be given placebo on Day 1 and Day 29.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CVnCoV Vaccine — Participants will receive an intramuscular injection by needle in the deltoid area.
  Other Names: CV07050101
  Arms: Dose Escalation CVnCoV
Drug: Placebo — Participants will receive an intramuscular injection by needle in the deltoid area.
  Arms: Dose Escalation Placebo

SUMMARY:
This study aims to evaluate the safety and reactogenicity profile after 1 and 2 dose administrations of CVnCoV at different dose levels.

DETAILED DESCRIPTION:
Funded by Coalition for Epidemic Preparedness Innovations (CEPI).

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria for all participants:

* Healthy male and female participants aged 18 to 60 years inclusive. Healthy participant is defined as an individual who is in good general health, not having any mental or physical disorder requiring regular or frequent medication.
* Expected to be compliant with protocol procedures and available for clinical follow-up through the last planned visit.
* Physical examination and laboratory results without clinically significant findings according to the Investigator's assessment.
* Body Mass Index (BMI) ≥18.0 and ≤30.0kg/m^2 (≥18.0 and ≤32.0kg/m2 for participants with SARS-CoV-2 positive serology).
* Females: At the time of enrollment, negative human chorionic gonadotropin (hCG) pregnancy test (serum) for women presumed to be of childbearing potential on the day of enrollment. On Day 1 (pre-vaccination): negative urine pregnancy test (hCG), (only required if the serum pregnancy test was performed more than 3 days before).
* Females of childbearing potential must use highly effective methods of birth control from 1 month before the first administration of the trial vaccine until 3 months following the last administration. The following methods of birth control are considered highly effective when used consistently and correctly:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal);
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable);
  * Intrauterine devices (IUDs);
  * Intrauterine hormone-releasing systems (IUSs);
  * Bilateral tubal occlusion;
  * Vasectomized partner;
  * Sexual abstinence (periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal are not acceptable).

Exclusion Criteria:

The following criterion applies to all open-label sentinel participants:

* Participants with SARS-CoV-2 positive serology as confirmed by testing at enrollment.

The following criteria apply to all participants, except those with SARS-CoV-2 positive serology:

* Participants considered at the Investigator's discretion to be at increased risk to acquire COVID-19 disease (including, but not limited to, health care workers with direct involvement in patient care or care of long-term care recipients).
* History of confirmed COVID-19 disease or known exposure to an individual with confirmed COVID-19 disease or SARS-CoV-2 infection within the past 2 weeks.

The following criteria apply to all participants:

* Use of any investigational or non-registered product (vaccine or drug) other than the trial vaccine within 28 days preceding the administration of the trial vaccine, or planned use during the trial period.
* Receipt of any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or planned receipt of any vaccine within 28 days of trial vaccine administration.
* Receipt of any investigational SARS-CoV-2 or other CoV vaccine prior to the administration of the trial vaccine.
* Any treatment with immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine or planned use during the trial, with the exception of topically-applied steroids. Corticosteroids used in the context of COVID-19 disease of participants with SARS CoV 2 positive serology are not exclusionary.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination, including known human immunodeficiency virus infection, hepatitis B virus infection and hepatitis C virus infection.
* History of a pIMD (potential immune-mediated disease).
* History of angioedema.
* Any known allergy, including allergy to any component of CVnCoV or aminoglycoside antibiotics. A history of hay fever or seasonal allergies (pollinosis) that does not require current treatment (e.g., anti-histamines) during the vaccination period (1 month before first vaccination until 1 month after last vaccination) is not exclusionary.
* History of or current alcohol and/or drug abuse.
* Participants who are active smokers, were active smokers within the last year (including any vaping in the last year) or have a total smoking history ≥10 pack years.
* Active or currently active SARS-CoV-2 infection as confirmed by reactive PCR within 3 days of first trial vaccine administration.
* History of confirmed SARS or MERS
* Administration of immunoglobulins (Igs) and/or any blood products within the 3 months preceding the administration of any dose of the trial vaccine.
* Presence or evidence of significant acute or chronic, medical or psychiatric illness. Significant medical or psychiatric illnesses include but are not limited to:

  * Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years.
  * Respiratory disease with clinically significant dyspnea in the last 5 years (except COVID-19 disease in participants with SARS-CoV-2 positive serology).
  * Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long- and short-acting beta agonists, theophylline, ipratropium, biologics.
  * Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease, history of stroke, peripheral artery disease, pulmonary embolism) or history of myocarditis or pericarditis as an adult.
  * Elevated blood pressure or hypertension, even if well-controlled.
  * Diabetes mellitus type 1 or 2.
  * History of any neurological disorders or seizures including Guillain-Barré syndrome, with the exception of febrile seizures during childhood.
  * Current or past malignancy, unless completely resolved without sequelae for >5 years.
* Foreseeable non-compliance with protocol as judged by the Investigator.
* For females: pregnancy or lactation.
* History of any anaphylactic reactions.
* Participants with impaired coagulation or any bleeding disorder in whom an IM injection or a blood draw is contraindicated.
* Participants employed by the Sponsor, Investigator or trial site, or relatives of research staff working on this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Universitair Ziekenhuis Ghent, Ghent, Belgium
- Germany (3):
  - Ludwig-Maximilians-Universität München, München, Bavaria
  - Medical University Hannover (MHH), Hanover
  - University Hospital Tübingen Institut für Tropenmedizin, Tübingen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed in Belgium and Germany between June 2020 and December 2021.
Pre-assignment Details: Of the 408 participants who were screened, 280 participants were enrolled.
Groups:
- Dose Escalation CVnCoV: 2 µg: Participants were vaccinated with CVnCoV at a dose of 2 µg on Day 1 and Day 29.
  Dose levels of 2, 4, 6, 8, 12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
- Dose Escalation CVnCoV: 4 µg: Participants were vaccinated with CVnCoV at a dose of 4 µg on Day 1 and Day 29.
  Dose levels of 2, 4, 6, 8, 12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
- Dose Escalation CVnCoV: 6 µg: Participants were vaccinated with CVnCoV at a dose of 6 µg on Day 1 and Day 29.
  Dose levels of 2, 4, 6, 8, 12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
- Dose Escalation CVnCoV: 8 µg: Participants were vaccinated with CVnCoV at a dose of 8 µg on Day 1 and Day 29.
  Dose levels of 2, 4, 6, 8, 12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
- Dose Escalation CVnCoV: 12 µg: Participants were vaccinated with CVnCoV at a dose of 12 µg on Day 1 and Day 29.
  Dose levels of 2, 4, 6, 8, 12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
- Dose Escalation CVnCoV: 16 µg: Participants were vaccinated with CVnCoV at a dose of 16 µg on Day 1 and Day 29.
  Dose levels of 2, 4, 6, 8, 12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
- Dose Escalation CVnCoV: 20 µg: Participants were vaccinated with CVnCoV at a dose of 20 µg on Day 1 and Day 29.
  Dose levels of 2, 4, 6, 8, 12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
- Dose Escalation Placebo: Participants were given placebo on Day 1 and Day 29.
  Placebo: Participants received an intramuscular injection by needle in the deltoid area.
Period: Overall Study
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Started | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Completed | 44 | 44 | 45 | 46 | 26 | 16 | 12 | 30
Not Completed | 3 | 4 | 3 | 3 | 2 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 3 | 2 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo | Total
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.48) | 39.1 (13.17) | 38.6 (12.74) | 38.9 (12.87) | 37.4 (13.51) | 37.4 (13.89) | 39.3 (12.11) | 40.1 (13.46) | 38.7 (12.85)
Age, Customized [Count of Participants; unit: Participants]
  18 - 40 years | 24 | 24 | 24 | 24 | 17 | 10 | 6 | 16 | 145
  41 - 60 years | 23 | 24 | 24 | 25 | 11 | 6 | 6 | 16 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 17 | 18 | 11 | 4 | 5 | 17 | 115
  Male | 27 | 25 | 31 | 31 | 17 | 12 | 7 | 15 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 44 | 48 | 46 | 49 | 27 | 16 | 11 | 32 | 273
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 43 | 48 | 44 | 47 | 28 | 16 | 12 | 31 | 269
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 34 | 30 | 38 | 45 | 25 | 12 | 8 | 26 | 218
  Belgium | 13 | 18 | 10 | 4 | 3 | 4 | 4 | 6 | 62
Baseline Immunestatus [Count of Participants; unit: Participants]
  Seropositive | 8 | 8 | 8 | 11 | 4 | 4 | 0 | 8 | 51
  Seronegative | 39 | 40 | 40 | 38 | 24 | 12 | 12 | 24 | 229

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 Adverse Reactions or Any Serious Adverse Event (SAE) Considered Related to Trial Vaccine Within at Least 24 Hours After the First Vaccination
Description: Grade 3 refers to the highest grading on the FDA toxicity scale where a higher grade indicates a worse outcome. An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
Time Frame: Up to 24 hours after vaccination on Day 1
Population: Only participants with available data were used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Any Grade 3 Adverse Reaction | 3 | 9 | 8 | 14 | 12 | 7 | 8 | 0
  Any Serious Adverse Event (SAE) Considered Related to Trial Vaccine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Grade 3 Adverse Reactions or Any Serious Adverse Event (SAE) Considered Related to Trial Vaccine Within at Least 60 Hours After the First Vaccination
Description: as for outcome 1
Time Frame: Up to 60 hours after vaccination on Day 1
Population: Only participants with available data were used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Any Grade 3 Adverse Reaction | 3 | 9 | 8 | 14 | 12 | 7 | 8 | 0
  Any Serious Adverse Event (SAE) Considered Related to Trial Vaccine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Local Adverse Events
Description: Reactogenicity was assessed daily via collection of solicited local AEs (injection site pain, redness, swelling, and itching) using paper diary cards.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Day 29 to 36)
Population: Only participants with available data were used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants | 32 | 43 | 38 | 41 | 26 | 16 | 11 | 5

4. Primary Outcome: Intensity of Solicited Local Adverse Events Per the FDA Toxicity Grading Scale
Description: Reactogenicity was assessed daily via collection of solicited local AEs (injection site pain, redness, swelling, and itching) using paper diary cards. Intensity of solicited local AEs and solicited systemic AEs were graded per the FDA Toxicity Grading Scale at Grades 1-3, where higher grades indicate a worse outcome.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: Per the statistical analysis plan for this endpoint, the overall number of participants analyzed includes all randomized participants to show the rate of grade 1, 2, and 3 events in the entire analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Placebo: Participants were be given placebo on Day 1 and Day 29.
  Placebo: Participants received an intramuscular injection by needle in the deltoid area.
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Grade 1 | 30 | 39 | 32 | 29 | 17 | 12 | 6 | 5
  Grade 2 | 2 | 3 | 5 | 11 | 9 | 4 | 5 | 0
  Grade 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0

5. Primary Outcome: Duration of Solicited Local Adverse Events
Description: Reactogenicity was assessed daily via collection of solicited local AEs (injection site pain, redness, swelling, and itching) using paper diary cards. Duration was calculated as consecutive days with a respective solicited AE regardless of the grade of the AE.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: Only participants who experienced solicited local AEs were used for this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 32 | 43 | 38 | 41 | 26 | 16 | 11 | 5
days | 1.8 (0.99) | 2.0 (0.84) | 2.3 (1.02) | 2.4 (1.44) | 2.6 (1.44) | 2.5 (0.82) | 3.0 (1.18) | 1.2 (0.45)

6. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events
Description: Reactogenicity was assessed daily via collection of solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) using paper diary cards.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: Only participants with available data were used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants | 29 | 45 | 44 | 45 | 28 | 16 | 12 | 19

7. Primary Outcome: Intensity of Solicited Systemic Adverse Events Per the FDA Toxicity Grading Scale
Description: Reactogenicity was assessed daily via collection of solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) using paper diary cards. Intensity of solicited local AEs and solicited systemic AEs were graded per the FDA Toxicity Grading Scale at Grades 1-3, where higher grades indicate a worse outcome.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Grade 1 | 21 | 22 | 20 | 11 | 1 | 2 | 0 | 15
  Grade 2 | 5 | 14 | 16 | 20 | 16 | 7 | 5 | 4
  Grade 3 | 3 | 9 | 8 | 14 | 11 | 7 | 7 | 0

8. Primary Outcome: Duration of Solicited Systemic Adverse Events
Description: Reactogenicity was assessed daily via collection of solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) using paper diary cards. Duration was calculated as consecutive days with a respective solicited AE regardless of the grade of the AE.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: Only participants who experienced solicited systemic AEs were used for this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 29 | 45 | 44 | 45 | 28 | 16 | 12 | 19
days | 3.1 (5.38) | 2.1 (1.15) | 2.4 (2.16) | 3.2 (2.40) | 3.6 (1.73) | 2.5 (0.73) | 3.4 (1.24) | 1.8 (0.96)

9. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events Considered Related to Trial Vaccine
Description: Reactogenicity was assessed daily via collection of solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) using paper diary cards. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to 7 days after vaccination (Days 1 to 8 and Days 29 to 36)
Population: Per the statistical analysis plan for this endpoint, the overall number of participants analyzed includes all randomized participants to show the number of participants with solicited adverse events considered related to trial vaccine in the entire analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants | 28 | 45 | 44 | 44 | 28 | 16 | 12 | 17

10. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Diaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants were contacted by phone to verify whether they had any health concerns since the last visit.
Time Frame: Up to 28 days after vaccination (Days 1 to 29 and Days 29 to 57)
Population: Only participants with available data were used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants | 26 | 32 | 29 | 31 | 23 | 13 | 11 | 16

11. Primary Outcome: Intensity of Unsolicited Adverse Events Assessed by the Investigator
Description: Diaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants were contacted by phone to verify whether they had any health concerns since the last visit. Participants were included only once, at the maximum severity. The Investigator made an assessment of intensity for each AE reported during the trial and assigned it to one of the following categories:
  * Mild: an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
  * Moderate: an event that caused sufficient discomfort to interfere with normal everyday activities.
  * Severe: an event that prevented normal everyday activities.
Time Frame: Up to 28 days after vaccination (Days 1 to 29 and Days 29 to 57)
Population: Per the statistical analysis plan for this endpoint, the overall number of participants analyzed includes all randomized participants to show the rate of mild, moderate, and severe adverse events in the entire analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Mild | 14 | 17 | 15 | 12 | 9 | 8 | 4 | 9
  Moderate | 10 | 13 | 10 | 17 | 10 | 5 | 2 | 6
  Severe | 2 | 2 | 4 | 2 | 4 | 0 | 5 | 1

12. Primary Outcome: Number of Participants With Unsolicited Adverse Events Considered Related to Trial Vaccine
Description: Diaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants were contacted by phone to verify whether they had any health concerns since the last visit. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to 28 days after vaccination (Days 1 to 29 and Days 29 to 57)
Population: Per the statistical analysis plan for this endpoint, the overall number of participants analyzed includes all randomized participants to show the number of participants with unsolicited adverse events considered related to trial vaccine in the entire analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation CVnCoV: 2 µg: Participants were vaccinated with CVnCoV at a dose of 2 µg on Day 1 and Day 29. Dose levels of 2, 4, 6, 8,12, 16, and 20 µg were evaluated.
  CVnCoV Vaccine: Participants received an intramuscular injection by needle in the deltoid area.
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants | 7 | 20 | 15 | 16 | 12 | 4 | 10 | 5

13. Primary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
Time Frame: Baseline to Day 393
Population: Only participants with available data were used in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 1

14. Primary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs) Considered Related to Trial Vaccine
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Baseline to Day 393
Population: Per the statistical analysis plan for this endpoint, the overall number of participants analyzed includes all randomized participants to show the number of participants with one or more SAEs considered related to trial vaccine in the entire analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With One or More Adverse Events of Special Interest (AESIs)
Description: The following events will be considered as AESIs: adverse events with a suspected immune-mediated etiology, COVID-19 disease and other adverse events relevant to SARS-CoV vaccine development or the target disease.
Time Frame: Day 1 to Day 393
Population: Only participants with available data were used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 47 | 48 | 48 | 49 | 28 | 16 | 12 | 28
Participants | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1

16. Secondary Outcome: Number of Participants Seroconverting for SARS-CoV-2 Spike Protein Antibodies
Description: Measured using Enzyme-Linked Immunosorbent Assay (ELISA). In participants who did not get exposed to SARS-CoV-2 before the trial or during the trial before the applicable sample was collected, as measured by ELISA to SARS-CoV-2 N-antigen, seroconversion is defined as an increase in titer in antibodies against SARS-CoV-2 spike protein versus baseline. In subjects seropositive for SARS-CoV-2 at baseline, seroconversion is defined as a 2-fold increase in titer in antibodies against SARS-CoV-2 spike protein versus baseline.
Time Frame: Day 8, Day 15, Day 29, Day 36, Day 43, Day 57, Day 120 and Day 211
Population: Participants who received at least 1 dose of trial vaccine and for whom the baseline blood sample and at least one additional blood sample are available for analysis (Immunogenicity Set).
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 46 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Day 8: number analyzed (Participants) | 46 | 48 | 45 | 46 | 28 | 16 | 12 | 32
  Day 8 | 18 | 17 | 19 | 19 | 9 | 8 | 6 | 12
  Day 15: number analyzed (Participants) | 45 | 47 | 44 | 45 | 25 | 16 | 12 | 32
  Day 15 | 23 | 22 | 23 | 28 | 14 | 11 | 7 | 8
  Day 29: number analyzed (Participants) | 45 | 46 | 45 | 46 | 27 | 16 | 12 | 31
  Day 29 | 26 | 27 | 27 | 29 | 16 | 15 | 11 | 9
  Day 36: number analyzed (Participants) | 45 | 44 | 43 | 45 | 28 | 16 | 12 | 30
  Day 36 | 42 | 44 | 39 | 39 | 27 | 16 | 12 | 17
  Day 43: number analyzed (Participants) | 43 | 44 | 45 | 45 | 28 | 16 | 12 | 29
  Day 43 | 42 | 44 | 43 | 44 | 26 | 16 | 12 | 12
  Day 57: number analyzed (Participants) | 42 | 44 | 47 | 47 | 26 | 16 | 11 | 31
  Day 57 | 38 | 42 | 38 | 43 | 24 | 16 | 11 | 7
  Day 120: number analyzed (Participants) | 45 | 47 | 48 | 46 | 27 | 16 | 12 | 30
  Day 120 | 29 | 39 | 31 | 34 | 26 | 15 | 12 | 10
  Day 211: number analyzed (Participants) | 43 | 42 | 43 | 44 | 26 | 16 | 11 | 29
  Day 211 | 23 | 31 | 22 | 27 | 24 | 16 | 10 | 8

17. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum SARS-CoV-2 Spike Protein Antibodies
Description: Measured using Enzyme-Linked Immunosorbent Assay (ELISA).
Time Frame: Day 8, Day 15, Day 29, Day 36, Day 43, Day 57, Day 120 and Day 211
Population: The Immunogenicity Set including only a subset of participants receiving 2 doses and who did not get exposed to SARS-CoV-2 before the trial, or during the trial before the applicable sample was collected, as measured by ELISA to SARS-CoV-2 N-antigen.
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 35 | 23 | 12 | 12 | 22
titers
  Day 8: number analyzed (Participants) | 36 | 37 | 34 | 32 | 23 | 12 | 12 | 22
  Day 8 | 133.655 (3.2545) | 147.911 (3.9771) | 236.879 (3.7524) | 126.603 (2.9179) | 154.168 (5.4433) | 75.715 (1.8549) | 251.617 (6.1263) | 157.993 (4.5998)
  Day 15: number analyzed (Participants) | 36 | 37 | 33 | 31 | 20 | 12 | 12 | 22
  Day 15 | 171.645 (2.8681) | 174.350 (3.5613) | 265.287 (3.6827) | 191.152 (2.4129) | 288.123 (6.6294) | 134.706 (2.8976) | 310.262 (6.7709) | 130.610 (4.3417)
  Day 29: number analyzed (Participants) | 36 | 37 | 37 | 35 | 23 | 11 | 12 | 22
  Day 29 | 173.625 (2.7202) | 216.617 (3.7230) | 284.084 (3.0997) | 210.045 (2.6297) | 253.696 (3.8848) | 415.167 (2.3220) | 497.175 (4.5434) | 129.860 (3.9097)
  Day 36: number analyzed (Participants) | 36 | 34 | 34 | 34 | 23 | 11 | 12 | 21
  Day 36 | 664.889 (2.9730) | 1700.053 (2.8334) | 1111.904 (2.8305) | 1254.241 (2.9320) | 1617.127 (3.2917) | 1163.062 (2.3845) | 1837.995 (3.4748) | 192.185 (3.8983)
  Day 43: number analyzed (Participants) | 34 | 33 | 36 | 34 | 23 | 11 | 12 | 20
  Day 43 | 1627.741 (2.6501) | 2375.689 (2.3220) | 2721.933 (2.7489) | 3052.067 (2.1718) | 3955.571 (3.3468) | 1815.393 (2.2767) | 6128.616 (2.8347) | 111.508 (3.9442)
  Day 57: number analyzed (Participants) | 33 | 34 | 36 | 34 | 21 | 11 | 11 | 21
  Day 57 | 1013.096 (2.8774) | 1845.542 (2.6503) | 1402.290 (2.3704) | 1591.849 (2.3855) | 2008.570 (2.6719) | 807.740 (2.2712) | 4793.501 (2.8151) | 108.232 (3.7280)
  Day 120: number analyzed (Participants) | 36 | 36 | 37 | 33 | 22 | 11 | 11 | 22
  Day 120 | 301.870 (4.3641) | 792.188 (2.2970) | 421.869 (3.3192) | 360.492 (2.4772) | 807.498 (2.9110) | 687.391 (3.4095) | 1100.769 (2.7710) | 99.688 (2.9239)
  Day 211: number analyzed (Participants) | 35 | 31 | 33 | 31 | 22 | 11 | 10 | 21
  Day 211 | 195.059 (3.0680) | 330.530 (2.8422) | 317.495 (4.2611) | 175.809 (2.3936) | 623.730 (2.8041) | 408.985 (2.0742) | 1027.909 (4.3847) | 84.518 (2.8642)

18. Secondary Outcome: Number of Participants Seroconverting for SARS-CoV-2 Spike Protein Receptor-Binding Domain (RBD) Antibodies
Description: Measured using Enzyme-Linked Immunosorbent Assay (ELISA). In participants who did not get exposed to SARS-CoV-2 before the trial or during the trial before the applicable sample was collected, as measured by ELISA to SARS-CoV-2 N-antigen, seroconversion is defined as an increase in titer in antibodies against SARS-CoV-2 spike RBD protein versus baseline. In subjects seropositive for SARS-CoV-2 at baseline, seroconversion is defined as a 2-fold increase in titer in antibodies against SARS-CoV-2 spike RBD protein versus baseline.
Time Frame: Day 8, Day 15, Day 29, Day 36, Day 43, Day 57, Day 120 and Day 211
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 46 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Day 8: number analyzed (Participants) | 46 | 48 | 45 | 46 | 28 | 16 | 12 | 32
  Day 8 | 8 | 8 | 8 | 13 | 4 | 5 | 1 | 7
  Day 15: number analyzed (Participants) | 45 | 47 | 44 | 45 | 25 | 16 | 12 | 32
  Day 15 | 8 | 8 | 10 | 10 | 4 | 5 | 1 | 5
  Day 29: number analyzed (Participants) | 45 | 46 | 45 | 46 | 27 | 16 | 12 | 31
  Day 29 | 9 | 11 | 9 | 12 | 7 | 6 | 2 | 4
  Day 36: number analyzed (Participants) | 45 | 44 | 43 | 45 | 28 | 16 | 12 | 30
  Day 36 | 20 | 30 | 26 | 34 | 21 | 14 | 8 | 3
  Day 43: number analyzed (Participants) | 43 | 44 | 45 | 45 | 28 | 16 | 12 | 29
  Day 43 | 31 | 37 | 37 | 43 | 26 | 16 | 12 | 2
  Day 57: number analyzed (Participants) | 42 | 44 | 47 | 49 | 26 | 16 | 11 | 31
  Day 57 | 23 | 32 | 33 | 40 | 23 | 16 | 11 | 2
  Day 120: number analyzed (Participants) | 45 | 47 | 48 | 46 | 27 | 16 | 12 | 30
  Day 120 | 13 | 22 | 24 | 34 | 20 | 13 | 11 | 3
  Day 211: number analyzed (Participants) | 43 | 42 | 43 | 44 | 26 | 16 | 11 | 29
  Day 211 | 7 | 13 | 16 | 17 | 17 | 8 | 9 | 1

19. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum SARS-CoV-2 Spike Protein Receptor-Binding Domain (RBD) Antibodies
Description: Measured using Enzyme-Linked Immunosorbent Assay (ELISA).
Time Frame: Day 8, Day 15, Day 29, Day 36, Day 43, Day 57, Day 120 and Day 211
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 35 | 23 | 12 | 12 | 22
titers
  Day 8: number analyzed (Participants) | 36 | 37 | 34 | 32 | 23 | 12 | 12 | 22
  Day 8 | 50.000 (1.0000) | 50.000 (1.0000) | 50.000 (1.0000) | 58.735 (1.5490) | 50.000 (1.0000) | 69.659 (2.9999) | 72.203 (3.5712) | 54.509 (1.3290)
  Day 15: number analyzed (Participants) | 36 | 37 | 33 | 31 | 20 | 12 | 12 | 22
  Day 15 | 50.000 (1.0000) | 50.000 (1.0000) | 55.894 (1.6444) | 53.520 (1.3017) | 50.000 (1.0000) | 68.942 (3.0430) | 74.942 (4.0629) | 52.644 (1.2734)
  Day 29: number analyzed (Participants) | 36 | 37 | 37 | 35 | 23 | 11 | 12 | 22
  Day 29 | 51.515 (1.1962) | 55.237 (1.4574) | 53.447 (1.5000) | 52.773 (1.2523) | 60.458 (1.5674) | 74.346 (2.7022) | 89.597 (4.1779) | 50.000 (1.0000)
  Day 36: number analyzed (Participants) | 36 | 34 | 34 | 34 | 23 | 11 | 12 | 21
  Day 36 | 92.943 (2.4539) | 201.936 (4.2892) | 144.011 (3.1421) | 255.615 (3.5880) | 351.489 (4.7386) | 321.393 (3.2174) | 388.660 (6.5376) | 54.303 (1.4598)
  Day 43: number analyzed (Participants) | 34 | 33 | 36 | 34 | 23 | 11 | 12 | 20
  Day 43 | 215.648 (3.3361) | 510.141 (4.0840) | 418.085 (3.9185) | 884.327 (3.5980) | 1401.175 (3.7419) | 1280.261 (2.6560) | 2035.914 (3.3154) | 54.694 (1.4938)
  Day 57: number analyzed (Participants) | 33 | 34 | 36 | 34 | 21 | 11 | 11 | 21
  Day 57 | 122.337 (3.0011) | 215.011 (3.5638) | 237.379 (3.7169) | 532.756 (3.3394) | 739.659 (3.9186) | 948.298 (2.7761) | 1516.255 (3.7810) | 50.000 (1.0000)
  Day 120: number analyzed (Participants) | 36 | 36 | 37 | 33 | 22 | 11 | 11 | 22
  Day 120 | 61.466 (1.7283) | 97.041 (2.5246) | 126.160 (3.6256) | 161.237 (2.5113) | 222.516 (3.4086) | 231.544 (2.8738) | 551.059 (3.7490) | 50.000 (1.0000)
  Day 211: number analyzed (Participants) | 35 | 31 | 33 | 31 | 22 | 11 | 10 | 21
  Day 211 | 50.000 (1.0000) | 73.596 (2.2529) | 102.077 (4.2320) | 70.541 (1.9584) | 208.484 (3.7448) | 139.858 (4.1588) | 390.307 (4.9577) | 50.000 (1.0000)

20. Secondary Outcome: Number of Participants Seroconverting for SARS-CoV-2 Neutralizing Antibodies
Description: Measured using an activity assay. In participants who did not get exposed to SARS-CoV-2 before the trial or during the trial before the applicable sample was collected, as measured by ELISA to SARS-CoV-2 N-antigen, seroconversion is defined as an increase in titer in SARS-CoV-2 neutralizing antibodies versus baseline. In participants seropositive for SARS-CoV-2 at baseline, seroconversion is defined as a 2-fold increase in titer in SARS-CoV-2 neutralizing antibodies versus baseline.
Time Frame: Day 8, Day 15, Day 29, Day 36, Day 43, Day 57, Day 120 and Day 211
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 46 | 48 | 48 | 49 | 28 | 16 | 12 | 32
Participants
  Day 8: number analyzed (Participants) | 46 | 48 | 45 | 46 | 28 | 16 | 12 | 32
  Day 8 | 7 | 8 | 8 | 12 | 4 | 4 | 1 | 3
  Day 15: number analyzed (Participants) | 45 | 47 | 44 | 45 | 25 | 16 | 12 | 32
  Day 15 | 8 | 7 | 9 | 21 | 4 | 4 | 2 | 4
  Day 29: number analyzed (Participants) | 45 | 46 | 45 | 46 | 27 | 16 | 12 | 31
  Day 29 | 8 | 9 | 9 | 19 | 3 | 5 | 2 | 2
  Day 36: number analyzed (Participants) | 45 | 44 | 43 | 45 | 28 | 16 | 12 | 30
  Day 36 | 24 | 28 | 29 | 35 | 23 | 12 | 9 | 4
  Day 43: number analyzed (Participants) | 43 | 44 | 45 | 45 | 28 | 16 | 12 | 29
  Day 43 | 34 | 35 | 36 | 39 | 25 | 15 | 10 | 4
  Day 57: number analyzed (Participants) | 42 | 44 | 47 | 47 | 26 | 16 | 11 | 31
  Day 57 | 26 | 24 | 28 | 45 | 22 | 14 | 9 | 4
  Day 120: number analyzed (Participants) | 45 | 47 | 48 | 46 | 27 | 16 | 12 | 30
  Day 120 | 16 | 18 | 22 | 28 | 16 | 10 | 11 | 2
  Day 211: number analyzed (Participants) | 43 | 42 | 43 | 44 | 26 | 16 | 11 | 29
  Day 211 | 13 | 14 | 22 | 19 | 7 | 5 | 5 | 2

21. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum SARS-CoV-2 Neutralizing Antibodies
Description: Measured using an activity assay.
Time Frame: Day 8, Day 15, Day 29, Day 36, Day 43, Day 57, Day 120 and Day 211
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 35 | 23 | 12 | 12 | 22
titers
  Day 8: number analyzed (Participants) | 36 | 37 | 34 | 32 | 23 | 12 | 12 | 22
  Day 8 | 5.000 (1.0000) | 5.000 (1.0000) | 5.000 (1.0000) | 5.221 (1.1859) | 5.000 (1.000) | 5.000 (1.0000) | 8.170 (5.4783) | 5.242 (1.2481)
  Day 15: number analyzed (Participants) | 36 | 37 | 33 | 31 | 20 | 12 | 12 | 22
  Day 15 | 5.000 (1.0000) | 5.000 (1.0000) | 5.106 (1.1282) | 8.269 (2.3683) | 5.000 (1.0000) | 5.000 (1.0000) | 9.715 (6.7304) | 5.000 (1.0000)
  Day 29: number analyzed (Participants) | 36 | 37 | 37 | 35 | 23 | 11 | 12 | 22
  Day 29 | 5.000 (1.0000) | 5.191 (1.2560) | 5.095 (1.1207) | 8.042 (2.3671) | 5.000 (1.0000) | 5.496 (1.3681) | 10.905 (7.3473) | 5.160 (1.1593)
  Day 36: number analyzed (Participants) | 36 | 34 | 34 | 34 | 23 | 11 | 12 | 21
  Day 36 | 12.240 (3.2214) | 17.340 (4.0855) | 13.577 (3.1691) | 26.336 (3.9767) | 22.224 (2.9539) | 14.142 (3.0248) | 38.860 (6.7690) | 5.430 (1.3051)
  Day 43: number analyzed (Participants) | 34 | 33 | 36 | 34 | 23 | 11 | 12 | 20
  Day 43 | 41.664 (5.0333) | 33.813 (4.0230) | 26.696 (4.2447) | 51.086 (3.5503) | 52.462 (3.4275) | 33.108 (3.2347) | 119.865 (6.8222) | 6.050 (1.8413)
  Day 57: number analyzed (Participants) | 33 | 34 | 36 | 34 | 21 | 11 | 11 | 21
  Day 57 | 13.419 (2.9626) | 11.892 (3.2240) | 13.348 (3.0155) | 49.044 (3.1527) | 24.786 (2.9671) | 28.284 (3.0577) | 96.647 (7.8329) | 5.612 (1.4462)
  Day 120: number analyzed (Participants) | 36 | 36 | 37 | 33 | 22 | 11 | 11 | 22
  Day 120 | 6.547 (1.6565) | 7.564 (2.0377) | 8.369 (2.2413) | 11.462 (2.2848) | 14.366 (3.1876) | 20.640 (5.0609) | 49.869 (4.5037) | 5.000 (1.0000)
  Day 211: number analyzed (Participants) | 35 | 31 | 33 | 31 | 22 | 11 | 10 | 21
  Day 211 | 7.001 (2.3126) | 9.247 (2.8688) | 11.107 (4.0813) | 8.086 (1.9730) | 6.234 (1.6616) | 5.325 (1.2324) | 11.487 (4.3194) | 5.000 (1.0000)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 393
Arm/Group | Dose Escalation CVnCoV: 2 µg | Dose Escalation CVnCoV: 4 µg | Dose Escalation CVnCoV: 6 µg | Dose Escalation CVnCoV: 8 µg | Dose Escalation CVnCoV: 12 µg | Dose Escalation CVnCoV: 16 µg | Dose Escalation CVnCoV: 20 µg | Dose Escalation Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/48 | 0/49 | 0/28 | 0/16 | 0/12 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/47 | 0/48 | 1/48 | 1/49 | 2/28 | 0/16 | 0/12 | 1/32
Other Adverse Events (participants affected / at risk) | 23/47 | 28/48 | 26/48 | 25/49 | 22/28 | 14/16 | 12/12 | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation CVnCoV: 2 µg (N=47) | Dose Escalation CVnCoV: 4 µg (N=48) | Dose Escalation CVnCoV: 6 µg (N=48) | Dose Escalation CVnCoV: 8 µg (N=49) | Dose Escalation CVnCoV: 12 µg (N=28) | Dose Escalation CVnCoV: 16 µg (N=16) | Dose Escalation CVnCoV: 20 µg (N=12) | Dose Escalation Placebo (N=32)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation CVnCoV: 2 µg (N=47) | Dose Escalation CVnCoV: 4 µg (N=48) | Dose Escalation CVnCoV: 6 µg (N=48) | Dose Escalation CVnCoV: 8 µg (N=49) | Dose Escalation CVnCoV: 12 µg (N=28) | Dose Escalation CVnCoV: 16 µg (N=16) | Dose Escalation CVnCoV: 20 µg (N=12) | Dose Escalation Placebo (N=32)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (10) | 7 (13) | 7 (10) | 4 (6) | 7 (13) | 5 (5) | 3 (3) | 3 (4)
Dizziness (Nervous system disorders) | 1 (2) | 6 (6) | 4 (5) | 4 (5) | 2 (5) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Morton's neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Feeling hot (General disorders) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (7) | 2 (2) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 2 (3) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Eccymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 3 (3) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmerorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04449276/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT04449276/SAP_001.pdf